CLINICAL TRIAL: NCT05983575
Title: A Study to Evaluate the Efficacy and Safety of LIPUS-Brain Transcranial Low-intensity Pulsed-wave Ultrasound Device in Patients With Early Alzheimer's Disease
Brief Title: A Pivotal Study of LIPUS-Brain in Patients With Early Alzheimer's Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sound Wave Innovation CO., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LB1101
Record Dates: First submitted 2023-07-18; First posted 2023-08-09 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease, Early Onset
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LIPUS-Brain (Experimental)
  Interventions: Device: LIPUS-Brain
- Placebo (Placebo Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: LIPUS-Brain — Transcranial low-power pulsed-wave ultrasound device
  Arms: LIPUS-Brain
Device: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized, double-blinded, placebo-controlled Phase 3 study comparing LIPUS-Brain transcranial low-intensity pulsed-wave ultrasound device to placebo in patients with Early Alzheimer's Disease. The primary objective of the study is to assess changes in ADAS-J-cog-14 scores from baseline to 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent to participate in the clinical trial from the patient and their legal representative.
* Mild AD or MCI due to AD patient aged greater than or equal to (>=) 50 and less than (<) 90 years, at the time of informed consent.
* Patients with the same partner/informant who meet all of the following conditions during the study period

  * Living with or in contact with the patient
  * It is possible to observe the patient's activities of daily living and physical condition.
  * Being able to be present at all times during the efficacy evaluation specified in this clinical trial
  * Person judged by an investigator to be able to manage administration of concomitant medications
* Patients who met the diagnostic criteria of Mild AD or MCI due to AD according to the NIA/AA 2018 diagnostic criteria at the time of informed consent and were diagnosed as positive by the amyloid PET imaging evaluation committee.
* Have a CDR global score of 0.5 (MCI due to AD) to 1.0 (Mild AD) at screening.
* Patients with her MMSE-J score >=20 at screening.
* No organic diseases such as symptomatic cerebral hemorrhage, symptomatic cerebral infarction, acute cerebral infarction, brain tumor, etc. within 48 weeks before obtaining informed consent or in head MRI images at screening, and in head MRA images, Patients evaluated by the imaging evaluation committee as not having severe stenosis/occlusion from the internal carotid artery to the middle cerebral artery.
* Patients who are receiving existing drug therapy for Mild AD or MCI due to AD and are not scheduled to change their medication within the past 4 weeks from obtaining consent and after obtaining consent.

Exclusion Criteria:

* Patients judged by the investigator that it is difficult to continue the study treatment for 20 minutes.
* Patients judged by the investigator to be difficult to perform an MRI examination.
* Patients with impaired consciousness with a GCS score of 12 or less at the time of enrollment.
* Patients who have had symptomatic cerebral infarction or cerebral hemorrhage within 12 weeks prior to enrollment.
* Patients with a modified Hachinski Ischemic Scale score of 5 or more at enrollment.
* Patients with Lewy body dementia and frontotemporal dementia.
* Patients judged by the investigator to be difficult to participate in the clinical trial due to severe mental illness
* Poorly controlled serious systemic disease (heart failure, liver failure, renal failure, vitamin B12 deficiency, hypothyroidism, etc.) that makes it difficult for the investigator to participate in the study judged patient.
* Patients with uncontrolled diabetic retinopathy (with active fundus hemorrhage).
* Patients who have malignant tumor as a complication or who have been treated for malignant tumor within 5 years from the time of enrollment (excluding cured resected carcinoma in situ).
* Patients who are or have a history of drug addiction or alcohol addiction.
* Patients with or with a history of epilepsy.
* Patients with implants such as coils, electrodes and stents in the skull.
* Patients within 5 years after brain surgery (including endovascular treatment).
* Patients who are pregnant or wish to become pregnant.
* Patients participating in other clinical studies (excluding non-interventional observational studies) or clinical trials.
* Patients who are otherwise judged to be ineligible by the investigator.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in ADAS-J-cog-14 scores from baseline to Week 72 | Performed at Week 72

SECONDARY OUTCOMES:
Changes in ADAS-J-cog-14 scores from baseline to Week 24 and 48 | Performed at Week 24 and 48
Changes in CDR-SB from baseline to Week 48 and 72 | Performed at Week 48 and 72
Changes in NPIQ-J scores from baseline to Week 24, 48 and 72 | Performed at Week 24, 48 and 72
Changes in J-ZBI scores from baseline to Week 24, 48 and 72 | Performed at Week 24, 48 and 72
Changes in WMS-R scores from baseline to Week 24, 48 and 72 | Performed at Week 24, 48 and 72
Changes in MMSE-J scores from baseline to Week 24, 48 and 72 | Performed at Week 24, 48 and 72
Changes in FAQ scores from baseline to Week 24, 48 and 72 | Performed at Week 24, 48 and 72
Changes in EQ-5D-5L scores from baseline to Week 24, 48 and 72 | Performed at Week 24, 48 and 72
Changes in ABC Dementia scale scores from baseline to Week 24, 48 and 72 | Performed at Week 24, 48 and 72
Changes in each 14 item of ADAS-J-cog-14 score from baseline to Week 24, 48 and 72 | Performed at Week 24, 48 and 72
Prevalence of responders at Week 24, 48, and 72 defined as those with no deterioration or even improvement in ADAS-J-cog-14 scores | Performed at Week 24, 48 and 72
Transition rate from MCI due to AD to AD at Week 72 | Performed at Week 72
Termination due to aggravation of dementia symptoms | Performed up to 96 weeks
  If medication needs to be started or changed, dementia is considered worsening.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Shimokawa, Study Director — Sound Wave Innovation CO., LTD.
Locations (19):
- Japan (19):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Center for Geriatrics and Gerontology, Ōbu, Aichi-ken
  - IUHW Narita Hospital, Narita, Chiba
  - Fukuoka Sanno Hospital, Fukuoka, Fukuoka
  - Imon Yukari Neurology Clinic, Hiroshima, Hiroshima
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Memory Clinic Toride, Toride, Ibaragi
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - KATAYAMA medical Clinic, Kurashiki, Okayama-ken
  - Kansai Medical University Hospital, Hirakata, Osaka
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - International University of Health and welfare Hospital, Nasushiobara, Tochigi
  - Juntendo University School of Medicine Juntendo Hospital, Bunkyō-Ku, Tokyo
  - Memory Clinic Ochanomizu, Bunkyō-Ku, Tokyo
  - The University of Tokyo Hospital, Bunkyō-Ku, Tokyo
  - Tokyo Metropolitan Geriatrics Hospital, Itabashi-ku, Tokyo
  - Tottori University Hospital, Yonago, Tottori

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shimokawa H, Akishita M, Asada T, Katayama S, Hattori Y, Yakushiji Y, Taki Y, Murai H, Boku Y, Tsujimoto M, Umegaki H, Ogawa T, Matsumoto S, Ono K, Imon Y, Tsunemi T, Iwata A, Hanajima R, Hisahara S, Uehara T, Ishiguro T, Nakaoku Y, Ishii K, Ishiki A, Nagai Y, Teramukai S, Ihara M, Fukushima M. Baseline characteristics of patients with early Alzheimer's disease enrolled in the pivotal trial of low-intensity pulsed ultrasound (LIPUS-AD). J Alzheimers Dis Rep. 2025 Dec 29;9:25424823251407541. doi: 10.1177/25424823251407541. eCollection 2025 Jan-Dec. PMID 41477670
- [Derived] Shimokawa H, Akishita M, Ihara M, Teramukai S, Ishiki A, Nagai Y, Fukushima M. Pivotal trial of low-intensity pulsed ultrasound therapy for early Alzheimer's disease: Rationale and design. J Alzheimers Dis Rep. 2025 Jan 13;9:25424823241312108. doi: 10.1177/25424823241312108. eCollection 2025 Jan-Dec. PMID 40034530